CLINICAL TRIAL: NCT05338060
Title: A Systems Approach to Immunotherapy Biomarker Identification Within the Postoperative Wound-Healing Microenvironment in Patients With Gastroesophageal Cancer
Acronym: BAISIC
Status: Completed | Type: Observational
Sponsor: Inova Health Care Services (Other)
Collaborators: George Mason University (Other)
Responsible Party: Sponsor
Other Study IDs: U21-05-4450
Record Dates: First submitted 2022-04-05; First posted 2022-04-20 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: GastroEsophageal Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — we will collect six to eight milliliters of fluid from surgical drains placed by the surgeon at the time of surgery to assist with wound healing. Samples will be collected at one and four to six days after surgery. One tube of blood will also be collected at both time points. The research will not include whole genome sequencing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: prospective collection of surgical exudates (SEs) — prospective collection of surgical exudates (SEs) from patients who are hospitalized for post-operative recovery from esophagectomy or gastrectomy for gastroesophageal cancer

SUMMARY:
The purpose of this research is to collect surgical drain fluid and blood from patients who have undergone surgery for gastric or esophageal cancer, and to analyze the fluid and blood using a variety of laboratory techniques for molecular markers capable of predicting response to immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing esophagectomy or gastrectomy for gastroesophageal cancer.
* Adult males and females at least 18 years of age
* Ability to complete testing in the protocol and attend study visits
* Able and willing to consent to protocol
* Adequate organ function Absolute Neutrophil Count (ANC) ≥1.5 x 103/μL Platelets ≥100 x 103/μL Hemoglobin >9.0 g/dL Total Bilirubin (</= 2.0 mg/dl at time of Y90 radioembolization) AST/ALT ≤5 x upper limit of normal Albumin >3 g/dL Creatinine ≤1.5 mg/dL

Exclusion Criteria:

* Female patients who are pregnant or breast-feeding
* Concomitant illness that would prevent adequate patient assessment or in the investigators' opinion pose an added risk for study participants.
* Life-threatening intercurrent illness
* Anticipated poor compliance
* Prisoners or subjects who are involuntarily incarcerated
* Persons with decisional incapacity/cognitive impairment
* Any history or evidence of severe illness or any other condition that would make the patient, in the opinion of the investigator unsuitable for the study
* Subject is enrolled in a separate interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult males and females at least 18 years of age undergoing esophagectomy or gastrectomy for gastroesophageal cancer
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Establishment of a workflow for collection of SEs from esophageal and gastric cancer patients. | 6 months
  to establish a workflow for collection of SEs from patients affected by esophageal and gastric cancer undergoing surgical resection.

SECONDARY OUTCOMES:
Assay characterization of SEs for Predictive and Prognostic Biomarkers to early vs. late/non-recurrence of malignancy. | 24 months
  SEs will be collected and characterized using different assays with the goal of generating hypotheses of potential predictive and prognostic biomarkers to early (<6 months) vs. late/non-recurrence of malignancy.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Wadlow, MD, Principal Investigator — Inova Schar Cancer Institute
Locations (1):
- Inova Schar Cancer Institute, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maleki Vareki S, Garrigos C, Duran I. Biomarkers of response to PD-1/PD-L1 inhibition. Crit Rev Oncol Hematol. 2017 Aug;116:116-124. doi: 10.1016/j.critrevonc.2017.06.001. Epub 2017 Jun 9. PMID 28693793
- [Background] Dholaria B, Hammond W, Shreders A, Lou Y. Emerging therapeutic agents for lung cancer. J Hematol Oncol. 2016 Dec 9;9(1):138. doi: 10.1186/s13045-016-0365-z. PMID 27938382
- [Background] Diggs LP, Hsueh EC. Utility of PD-L1 immunohistochemistry assays for predicting PD-1/PD-L1 inhibitor response. Biomark Res. 2017 Mar 15;5:12. doi: 10.1186/s40364-017-0093-8. eCollection 2017. PMID 28331612
- [Background] Grigg C, Rizvi NA. PD-L1 biomarker testing for non-small cell lung cancer: truth or fiction? J Immunother Cancer. 2016 Aug 16;4:48. doi: 10.1186/s40425-016-0153-x. eCollection 2016. PMID 27532023
- [Background] Sundaram GM, Quah S, Sampath P. Cancer: the dark side of wound healing. FEBS J. 2018 Dec;285(24):4516-4534. doi: 10.1111/febs.14586. Epub 2018 Jun 25. PMID 29905002
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Background] Fuse N, Nagahisa-Oku E, Doi T, Sasaki T, Nomura S, Kojima T, Yano T, Tahara M, Yoshino T, Ohtsu A. Effect of RECIST revision on classification of target lesions and overall response in advanced gastric cancer patients. Gastric Cancer. 2013 Jul;16(3):324-8. doi: 10.1007/s10120-012-0187-9. Epub 2012 Aug 22. PMID 22910898
- [Background] Schwartz LH, Colville JA, Ginsberg MS, Wang L, Mazumdar M, Kalaigian J, Hricak H, Ilson D, Schwartz GK. Measuring tumor response and shape change on CT: esophageal cancer as a paradigm. Ann Oncol. 2006 Jun;17(6):1018-23. doi: 10.1093/annonc/mdl058. Epub 2006 Apr 26. PMID 16641170
- [Background] Pierobon M, Wulfkuhle J, Liotta L, Petricoin E. Application of molecular technologies for phosphoproteomic analysis of clinical samples. Oncogene. 2015 Feb 12;34(7):805-14. doi: 10.1038/onc.2014.16. Epub 2014 Mar 10. PMID 24608425
- [Background] Baldelli E, Calvert V, Hodge A, VanMeter A, Petricoin EF 3rd, Pierobon M. Reverse Phase Protein Microarrays. Methods Mol Biol. 2017;1606:149-169. doi: 10.1007/978-1-4939-6990-6_11. PMID 28502000
- [Background] Aebersold R, Mann M. Mass spectrometry-based proteomics. Nature. 2003 Mar 13;422(6928):198-207. doi: 10.1038/nature01511. PMID 12634793
- [Background] Poste G. Bring on the biomarkers. Nature. 2011 Jan 13;469(7329):156-7. doi: 10.1038/469156a. No abstract available. PMID 21228852
- [Background] Gerszten RE, Accurso F, Bernard GR, Caprioli RM, Klee EW, Klee GG, Kullo I, Laguna TA, Roth FP, Sabatine M, Srinivas P, Wang TJ, Ware LB. Challenges in translating plasma proteomics from bench to bedside: update from the NHLBI Clinical Proteomics Programs. Am J Physiol Lung Cell Mol Physiol. 2008 Jul;295(1):L16-22. doi: 10.1152/ajplung.00044.2008. Epub 2008 May 2. PMID 18456800
- [Background] Prakash A, Rezai T, Krastins B, Sarracino D, Athanas M, Russo P, Zhang H, Tian Y, Li Y, Kulasingam V, Drabovich A, Smith CR, Batruch I, Oran PE, Fredolini C, Luchini A, Liotta L, Petricoin E, Diamandis EP, Chan DW, Nelson R, Lopez MF. Interlaboratory reproducibility of selective reaction monitoring assays using multiple upfront analyte enrichment strategies. J Proteome Res. 2012 Aug 3;11(8):3986-95. doi: 10.1021/pr300014s. Epub 2012 Jul 3. PMID 22639787
- [Background] Luchini A, Fredolini C, Espina BH, Meani F, Reeder A, Rucker S, Petricoin EF 3rd, Liotta LA. Nanoparticle technology: addressing the fundamental roadblocks to protein biomarker discovery. Curr Mol Med. 2010 Mar;10(2):133-41. doi: 10.2174/156652410790963268. PMID 20196732
- [Background] Fredolini C, Meani F, Luchini A, Zhou W, Russo P, Ross M, Patanarut A, Tamburro D, Gambara G, Ornstein D, Odicino F, Ragnoli M, Ravaggi A, Novelli F, Collura D, D'Urso L, Muto G, Belluco C, Pecorelli S, Liotta L, Petricoin EF 3rd. Investigation of the ovarian and prostate cancer peptidome for candidate early detection markers using a novel nanoparticle biomarker capture technology. AAPS J. 2010 Dec;12(4):504-18. doi: 10.1208/s12248-010-9211-3. Epub 2010 Jun 12. PMID 20549403
- [Background] Pin E, Sjoberg R, Andersson E, Hellstrom C, Olofsson J, Jernbom Falk A, Bergstrom S, Remnestal J, Just D, Nilsson P, Manberg A. Array-Based Profiling of Proteins and Autoantibody Repertoires in CSF. Methods Mol Biol. 2019;2044:303-318. doi: 10.1007/978-1-4939-9706-0_19. PMID 31432421
- [Background] Park CH, Lee JG, Lee AR, Eun CS, Han DS. Network construction of gastric microbiome and organization of microbial modules associated with gastric carcinogenesis. Sci Rep. 2019 Aug 27;9(1):12444. doi: 10.1038/s41598-019-48925-4. PMID 31455798
- [Background] Popper U, Rumpold H. Update ESMO: gastric and esophageal cancer. memo - Magazine of European Medical Oncology. 2021;14:180-3.
- [Result] Shitara K, Ozguroglu M, Bang YJ, Di Bartolomeo M, Mandala M, Ryu MH, Fornaro L, Olesinski T, Caglevic C, Chung HC, Muro K, Goekkurt E, Mansoor W, McDermott RS, Shacham-Shmueli E, Chen X, Mayo C, Kang SP, Ohtsu A, Fuchs CS; KEYNOTE-061 investigators. Pembrolizumab versus paclitaxel for previously treated, advanced gastric or gastro-oesophageal junction cancer (KEYNOTE-061): a randomised, open-label, controlled, phase 3 trial. Lancet. 2018 Jul 14;392(10142):123-133. doi: 10.1016/S0140-6736(18)31257-1. Epub 2018 Jun 4. PMID 29880231
- [Result] Kojima T, Shah MA, Muro K, Francois E, Adenis A, Hsu CH, Doi T, Moriwaki T, Kim SB, Lee SH, Bennouna J, Kato K, Shen L, Enzinger P, Qin SK, Ferreira P, Chen J, Girotto G, de la Fouchardiere C, Senellart H, Al-Rajabi R, Lordick F, Wang R, Suryawanshi S, Bhagia P, Kang SP, Metges JP; KEYNOTE-181 Investigators. Randomized Phase III KEYNOTE-181 Study of Pembrolizumab Versus Chemotherapy in Advanced Esophageal Cancer. J Clin Oncol. 2020 Dec 10;38(35):4138-4148. doi: 10.1200/JCO.20.01888. Epub 2020 Oct 7. PMID 33026938
- [Result] Kato K, Cho BC, Takahashi M, Okada M, Lin CY, Chin K, Kadowaki S, Ahn MJ, Hamamoto Y, Doki Y, Yen CC, Kubota Y, Kim SB, Hsu CH, Holtved E, Xynos I, Kodani M, Kitagawa Y. Nivolumab versus chemotherapy in patients with advanced oesophageal squamous cell carcinoma refractory or intolerant to previous chemotherapy (ATTRACTION-3): a multicentre, randomised, open-label, phase 3 trial. Lancet Oncol. 2019 Nov;20(11):1506-1517. doi: 10.1016/S1470-2045(19)30626-6. Epub 2019 Sep 30. PMID 31582355
- [Result] Moehler M, Shitara K, Garrido M, Salman P, Shen L, Wyrwicz L, et al. LBA6_PR Nivolumab (nivo) plus chemotherapy (chemo) versus chemo as first-line (1L) treatment for advanced gastric cancer/gastroesophageal junction cancer (GC/GEJC)/esophageal adenocarcinoma (EAC): First results of the CheckMate 649 study. Annals of Oncology. 2020;31:S1191.
- [Result] Kato K, Sun JM, Shah MA, Enzinger PC, Adenis A, Doi T, et al. LBA8_PR Pembrolizumab plus chemotherapy versus chemotherapy as first-line therapy in patients with advanced esophageal cancer: The phase 3 KEYNOTE-590 study. Annals of Oncology. 2020;31:S1192-S3.
- [Result] Kelly RJ, Ajani JA, Kuzdzal J, Zander T, Van Cutsem E, Piessen G, Mendez G, Feliciano J, Motoyama S, Lievre A, Uronis H, Elimova E, Grootscholten C, Geboes K, Zafar S, Snow S, Ko AH, Feeney K, Schenker M, Kocon P, Zhang J, Zhu L, Lei M, Singh P, Kondo K, Cleary JM, Moehler M; CheckMate 577 Investigators. Adjuvant Nivolumab in Resected Esophageal or Gastroesophageal Junction Cancer. N Engl J Med. 2021 Apr 1;384(13):1191-1203. doi: 10.1056/NEJMoa2032125. Erratum In: N Engl J Med. 2023 Feb 16;388(7):672. doi: 10.1056/NEJMx220014. PMID 33789008